CLINICAL TRIAL: NCT02249429
Title: Open-Label, Non Randomized Phase 2 Study With Safety Run-In Evaluating Efficacy and Safety of PQR309 in Patients With Relapsed or Refractory Lymphoma
Brief Title: Open-Label, Non Randomized Phase 2 Study With Safety Run-In
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PIQUR Therapeutics AG (Industry)
Collaborators: University College London Hospitals (Other); Churchill Hospital (Other); Royal Marsden NHS Foundation Trust (Other); University of Haifa (Other); Weill Medical College of Cornell University (Other); Institut Curie (Other); University Clinical Center, Sarajevo (Unknown); Clinical Center Kragujevac (Other); Clinical Center Nis, Nis (Unknown); Institute for Oncology and Radiology Serbia, Belgrade (Unknown); University Clinical Centre of Republic of Srpska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQR309-002
Record Dates: First submitted 2014-09-08; First posted 2014-09-25 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Lymphoma, Malignant
Keywords: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Phosphatidylinositol 3-Kinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- bimiralisib (PQR309) (Experimental)
  Interventions: Drug: bimiralisib

INTERVENTIONS:
Drug: bimiralisib — 60 mg or 80 mg bimiralisib per oral (p.o.) once daily or intermittent dosing (120mg,140mg and 160mg) until unacceptable AE, disease progression, patient's request for withdrawal, investigator judgement or death - whichever comes first.
  Other Names: PQR309; PI3K Inhibitor (phosphatidylinositol 3-kinase)

SUMMARY:
The main goal of this study is to determine the Maximum Tolerated Dose (MTD) and the Recommended Phase II Dose (RP2D) as well as preliminary antitumor activity of bimiralisib (PQR309) administered orally, as once daily capsules continuously and on intermittent schedule in patients with relapsed or refractory lymphomas.

DETAILED DESCRIPTION:
Open-label, non-randomized, multicentre phase 2 study with a safety run-in evaluating efficacy and safety of bimiralisib (PQR309) in patients with relapsed or refractory lymphoma.

The maximum tolerated dose (MTD) of bimiralisib in patients with advanced solid tumors was defined as 80 mg once daily given continuously (q.d. schedule) in a previous phase 1 study. The safety run-in of this study will follow a modified 3 + 3 design to evaluate the safety of 60 and 80 mg bimiralisib in patients with relapsed or refractory lymphoma administered p.o. once daily during a DLT (dose-limiting toxicity) period of 28 days.

In the safety run-in, three patients will be treated at 60 mg bimiralisib for 28 days. Enrollment and treatment of all three patients may occur simultaneously as 80 mg bimiralisib p.o. qd was established as the MTD in solid tumors. Unless a DLT is observed in any of the three patients during the first 28 days of treatment, the investigators and the sponsor will decide to escalate the dose to 80 mg. Intermittent dosing schedules may be evaluated if, based on the overall evaluation of all the clinical and PK (pharmacokinetic) data from this and other studies with bimiralisib, data emerge during step 1 of the phase 2 expansion in this study, indicating that daily dosing of bimiralisib is not adequately tolerated or inefficacious.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis* of relapsed or refractory lymphoma, received at least two prior lines of therapy including immuno-chemotherapy. Patients with relapsed Chronic Lymphoid Leukemia (CLL) are eligible if they have received one or more prior lines of any approved standard therapy. * archival biopsies may be used if obtained up to a year prior to enrollment; re-biopsy is strongly recommended if last biopsy was obtained more than a year ago.
2. Only for patients in the Phase 2 part: At least one measurable nodal or extra-nodal lesion defined as follows: Clearly measurable (i.e. well-defined boundaries) in at least two perpendicular dimensions on imaging scan with > 1.5 cm in longest transverse diameter.
3. Age ≥ 18 years
4. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1 (See Appendix 2).
5. Adequate organ system functions defined as:

   1. Absolute neutrophil count (ANC) ≥1.0x109/l
   2. Platelets ≥ 75x109/l
   3. Haemoglobin ≥ 85g/L
   4. Adequate hepatic function, defined as Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) and Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN (or ALT/AST ≤ 5 times ULN in patients with liver involvement)
   5. Adequate renal function, defined as serum creatinine ≤ 1.5 times ULN
   6. Fasting glucose < 7.0 mmol/L; Glycated haemoglobin (HbA1c) < 6.4%
6. Ability and willingness to swallow and retain oral medication.
7. Willingness and ability to comply with the trial procedures
8. Female and male patients with reproductive potential must agree to use effective contraception from screening until 90 days after discontinuation of PQR309
9. Signed informed consent

Exclusion Criteria:

Any of the following conditions precludes enrollment of a patient:

1. Immunosuppression due to:

   * Allogeneic hematopoietic stem cell transplant (HSCT)
   * Any immune-suppressive therapy within 4 weeks prior to trial treatment start
   * Known HIV infection
2. Autologous stem cell transplant within 3 months prior to trial treatment start.
3. Concomitant anticancer therapy (e.g. chemotherapy, radiotherapy, hormonal therapy, immunotherapy, biological response modifier, signal transduction inhibitors).
4. Concomitant treatment with medicinal products that increase the pH (reduce acidity) of the upper gastrointestinal tract, including, but not limited to, proton-pump inhibitors (e.g. omeprazole), H2-antagonists (e.g. ranitidine) and antacids. Patients may be enrolled in the study after a wash-out period sufficient to terminate their effect.
5. Use of any investigational drug within 21 days prior to trial treatment start.
6. Patients who experienced National Cancer Institute (NCI) Common Terminology Criteria For Adverse Events (CTCAE) ≥ Grade 3 on PI3K/mTOR inhibitors
7. Any major surgery, chemotherapy or immunotherapy within 21 days prior to trial treatment start.
8. Symptomatic or progressing Central nervous system (CNS) involvement. Exception: Patients with meningeal involvement can be included upon discussion between the sponsor and the investigator.
9. Persisting toxicities NCI CTCAE ≥2 related to prior anticancer therapy
10. Presence of gastrointestinal disease or any other condition that could interfere significantly with the absorption of the study drug.
11. Severe/unstable angina, myocardial infarction or coronary artery bypass within the last 3 years prior to trial treatment start, symptomatic congestive heart failure New York Heart Association (NYHA) Class 3 or 4, hypertension BP>150/100mmHg
12. A serious active infection at the time of treatment, or another serious underlying medical condition that could impair the ability of the patient to receive treatment.
13. Lack of appropriate contraceptive measures (male and female)
14. Pregnant or lactating women
15. Known HIV infection
16. Significant medical conditions which could jeopardize compliance with the protocol.
17. Uncontrolled diabetes mellitus; patients with controlled diabetes may be enrolled (see fasting glucose and HbA1c levels in inclusion criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Change of Tumor Response Criteria in lymphoma patients During Treatment with PQR309 in patients with relapsed or refractory lymphoma according to Cheston Criteria (5) | 28 day prior to first treatment (baseline), during treatment every 8 weeks during 6 months and every 6 months afterwards up to 1 year)
  Radiological lymphoma Evaluation (CT or other indicated according to institutional standard practice), clinical examination and bone marrow biopsy

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAE) and severity of all adverse events (AEs) | Before treatment on Day -1,-2 and during treatment on Day 1,2,8,15,22,36,50, at the end of treatment up to 1 year and 30 days after last dose
  Continuous dosing and intermittent dosing
Change of pulse rate | Before treatment on Day -1,-2 and during treatment on Day 1,2,8,15,22,36,50, at the end of treatment up to 1 year and 30 days after last dose
  Continuous dosing and intermittent dosing
Change in blood pressure | Before treatment on Day -1,-2 and during treatment on Day 1,2,8,15,22,36,50, subsequently every 4 weeks up to 1 year, at the end of treatment up to 1 year and 30 days after last dose
  Continuous dosing and intermittent dosing
Change in body temperature | Before treatment on Day -1,-2 and during treatment on Day 1,2,8,15,22,36,50, subsequently every 4 weeks up to 1 year, at the end of treatment up to 1 year and 30 days after last dose
  Continuous dosing and intermittent dosing
Change in ECOG (Eastern Cooperative Oncology Group) Performance status | Before treatment on Day -1,-2 and during treatment on Day 1,2,8,15,22,36,50, subsequently every 4 weeks up to 1 year, at the end of treatment up to 1 year and 30 days after last dose
  Continuous dosing and intermittent dosing
Change in body weight | Before treatment on Day -1,-2 and during treatment on Day 1,2,8,15,22,36,50, subsequently every 4 weeks up to 1 year, at the end of treatment up to 1 year and 30 days after last dose
  Continuous dosing and intermittent dosing
Change in haematology | Before treatment on Day -1,-2 and during treatment on Day 1,2,8,15,22,36,50, subsequently every 4 weeks up to 1 year, at the end of treatment up to 1 year and 30 days after last dose
  Continuous dosing and intermittent dosing
Change in blood chemistry | Before treatment on Day -1 and during treatment on Day 1,22,50, subsequently every 4 weeks up to 1 year, at the end of treatment up to 1 year
  Continuous dosing and intermittent dosing
Change in ECG (electrocardiogram) | Before treatment on Day -1 and during treatment on Day 1,22,50, subsequently every 4 weeks up to 1 year, at the end of treatment up to 1 year
  Continuous dosing and intermittent dosing
Change of urine analysis | Before treatment on Day -1 and during treatment on Day 1,22,50, subsequently every 4 weeks up to 1 year, at the end of treatment up to 1 year
  Continuous dosing and intermittent dosing
Change in HbA1c | Before treatment on Day -1 and during treatment on Day 1,22,50, subsequently every 4 weeks up to 1 year, at the end of treatment up to 1 year
  Continuous dosing and intermittent dosing
Change in tmax | During treatment on Day 1,2, 8,15 22, 50
  Continuous dosing and intermittent dosing
Change in Cmax | During treatment on Day 1,2, 8,15 22, 50
  Continuous dosing and intermittent dosing
Change in AUC 0-24 | During treatment on Day 1,2, 8,15 22, 50
  Continuous dosing and intermittent dosing
Change in AUClast | During treatment on Day 1,2, 8,15 22, 50
  Continuous dosing and intermittent dosing
Change in AUC0-∞, | During treatment on Day 1,2, 8,15 22, 50
  Continuous dosing and intermittent dosing
Change in t1/2 | During treatment on Day 1,2, 8,15 22, 50
  Continuous dosing and intermittent dosing
Change in RAC | During treatment on Day 1,2, 8,15 22, 50
  Continuous dosing and intermittent dosing

OTHER OUTCOMES:
Change in insulin/ C-Peptide/ glucose | During treatment on Day 1,2, 8,15 22, 50
  Continuous dosing and intermittent dosing

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Popat, Principal Investigator — Univeristy College London; David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust; Paul Fields, Principal Investigator — Guy's Hospital; Graham Collins, Principal Investigator — Churchill Hospital; Netanel Horowitz, Principal Investigator — University of Haifa; Giulino Roth, Principal Investigator — Weill Cornell Medicine New York; Carole Soussain, Principal Investigator — Curie Institute; Sinisa Radulovic, Principal Investigator — Institute for Oncology and Radiology Serbia; Ivan Tijanic, Principal Investigator — Clinical Center Nis; Nebojsa Andjelkovic, Principal Investigator — Clinical Center Kragujevac; Sabrina Kurtovic, Principal Investigator — University Clinical Center, Sarajevo; Danijela Mandic, Principal Investigator — University Clinical Centre of Republic of Srpska
Locations (12):
- Weill Cornell Medicine, New York, New York, United States
- Bosnia and Herzegovina (2):
  - University Clinical Center Republic of Srpska, Banja Luka
  - University Clinical Center Sarajevo, Sarajevo
- Insitute Curie, Saint-Cloud, Paris, France
- Univeristy Hospital Haifa, Haifa, Israel
- Serbia (3):
  - Institute for Oncology and radiology of Serbia, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
- United Kingdom (4):
  - Guy's Hospital, London
  - Royal Marsden NHS Foundation Trust, London
  - University College Hospital London, London
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No